CLINICAL TRIAL: NCT01589237
Title: An Open Label, 52-week, Safety and Tolerability Extension to a Randomized, Double-blind, Placebo Controlled Study of LCQ908 in Subjects With Familial Chylomicronemia Syndrome.
Brief Title: Extension to a Randomized, Double-blind, Placebo Controlled Study of LCQ908 in Subjects With Familial Chylomicronemia Syndrome.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Interim analysis suggested that size of benefit anticipated from continued participation of patients in Part B no longer supported trial extension beyond Part A
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLCQ908B2305; 2012-000802-32 (EudraCT Number)
Record Dates: First submitted 2012-04-27; First posted 2012-05-01 (Estimated); Results first posted 2016-11-15 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-09

CONDITIONS: Familial Chylomicronemia Syndrome (FCS) (HLP Type I)
Keywords: Familial Chylomicronemia Syndrome (FCS) (HLP type I); LCQ908
MeSH Terms: conditions — Familial hyperchylomicronemia syndrome | interventions — pradigastat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LCQ908 (Experimental): Patients initiated at 10 mg/day. After at least 8 weeks of treatment with a dose, optional up-titration to the next possible dose will be allowed. One down titration allowed from the highest dose attained.
  Interventions: Drug: LCQ908

INTERVENTIONS:
Drug: LCQ908

SUMMARY:
This study was to determine long-term safety and tolerability, and continued efficacy in lowering triglycerides of LCQ908 in subjects with Familial Chylomicronemia Syndrome (FCS) (HLP type I).

DETAILED DESCRIPTION:
This study was an 52 weeks open label extension starting at the lowest treatment dose used in CLCQ908B2302/NCT01514461 (i.e., 10 mg) with optional up-titrations, to evaluate the overall long-term safety and tolerability of LCQ908 in patients with Familial Chylomicronemia Syndrome, who either discontinued from the CLCQ908B2302/NCT01514461 study (due to tolerability issues) or completed the CLCQ908B2302/NCT01514461 study after 52 weeks. In addition, patients who had previously completed study CLCQ908A2212/NCT01146522 were eligible to participate.

Following Protocol amendment 2, the original 52 week duration of this study (CLCQ908B2305) became Part A of LCQ908B2305 and a 78 week extension became Part B. However, following Protocol amendment 3, Part B was ended at the same time as the last patient of Part A completed 52 weeks. The reason for termination of Part B was the findings from the December 2014 interim analysis which suggested that the size of benefit that was anticipated from continued participation of patients in the 18 month extension trial (Part B) no longer supported trial extension beyond Part A.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before any assessment is performed.
2. Subjects that either discontinue prematurely or complete the CLCQ908B2302 study after 52 weeks or FCS subjects who have previously completed study CLCQ908A2212.

Exclusion Criteria:

1. Subjects discontinued from the CLCQ908B2302 study for serious, potentially study drug related adverse events.
2. Subjects from the CLCQ908B2302 study who have developed any other contraindication to participation (for example, renal failure)
3. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
4. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
5. Subjects with type 1 diabetes mellitus or type 2 diabetes mellitus if HbA1C is ≥ 8.5%.
6. Treatment with fish oil preparations within 4 weeks prior to randomization.
7. Treatment with bile acid binding resins (i.e., colesevelam, etc) within 4 weeks prior to randomization.
8. Treatment with fibrates within 8 weeks prior to randomization. Washout may occur following screening if required.
9. Glybera [alipogene tiparvovec (AAV1-LPLS447X )] gene therapy exposure within the two years prior to screening.
10. eGFR <45 ml/min/1.73m2 or history of chronic renal disease.

Other protocol defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-02; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- Novartis Investigative Site, Seatlle, Washington, United States
- Canada (3):
  - Novartis Investigative Site, Chicoutimi, Quebec
  - Novartis Investigative Site, Ste-Foy, Quebec
  - Novartis Investigative Site, Ouest-Montreal
- France (2):
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
- Novartis Investigative Site, Hamburg, Germany
- Novartis Investigative Site, Meibergdreef 9, Netherlands
- Novartis Investigative Site, Cape Town, South Africa
- Novartis Investigative Site, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 100% patients who completed the screening phase were enrolled in the study.
Groups:
- Placebo of Pradigastat (LCQ908) Regimen: Part A: Patients who were randomized to placebo in study CLCQ908B2302/NCT01514461. In current study, patients initiated at 10 mg/day. After at least 8 weeks of treatment with a dose, optional up-titration to the next possible dose was allowed. One down titration allowed from the highest dose attained.
  Part B: Patients who consented to take part in the Part B continued their treatment at the same dose as they took when they completed Part A. LCQ908 treatment could be titrated (within the dose range 10 mg to 40 mg) at the investigators discretion and based on individual patients' tolerance and safety profile.
- 20 mg Pradigastat (LCQ908) Regimen: Part A: Patients who were randomized to LCQ908 20 mg in study CLCQ908B2302/NCT01514461. In current study, patients initiated at LCQ908 10 mg/day. After at least 8 weeks of treatment with a dose, optional up-titration to the next possible dose was allowed. One down titration allowed from the highest dose attained.
  Part B: Patients who consented to take part in the Part B continued their treatment at the same dose as they took when they completed Part A. LCQ908 treatment could be titrated (within the dose range 10 mg to 40 mg) at the investigators discretion and based on individual patients' tolerance and safety profile.
- 40 mg Pradigastat (LCQ908) Regimen: Part A: Patients who were randomized to LCQ908 40 mg in study CLCQ908B2302/NCT01514461. In current study, patients initiated at LCQ908 10 mg/day. After at least 8 weeks of treatment with a dose, optional up-titration to the next possible dose was allowed. One down titration allowed from the highest dose attained.
  Part B: Part B: Patients who consented to take part in the Part B continued their treatment at the same dose as they took when they completed Part A. LCQ908 treatment could be titrated (within the dose range 10 mg to 40 mg) at the investigators discretion and based on individual patients' tolerance and safety profile.
- Pradigastat (LCQ908) Regimen- From Study A2212: Part A: Patients who were randomized to LCQ908 in study CLCQ908A2212/NCT01146522. In current study, patients initiated at LCQ908 10 mg/day. After at least 8 weeks of treatment with a dose, optional up-titration to the next possible dose was allowed. One down titration allowed from the highest dose attained.
  Part B: Patients who consented to take part in the Part B continued their treatment at the same dose as they took when they completed Part A. LCQ908 treatment could be titrated (within the dose range 10 mg to 40 mg) at the investigators discretion and based on individual patients' tolerance and safety profile.
Period: Part A (52 Weeks)
Arm/Group | Placebo of Pradigastat (LCQ908) Regimen | 20 mg Pradigastat (LCQ908) Regimen | 40 mg Pradigastat (LCQ908) Regimen | Pradigastat (LCQ908) Regimen- From Study A2212
Started | 11 ("Started" = Full analysis set/safety set) | 12 | 10 | 5
Completed | 9 | 9 | 8 | 5
Not Completed | 2 | 3 | 2 | 0
Not completed — Subject/guardian decision | 2 | 3 | 2 | 0
Period: Part B (Planned for 78 Week-terminated)
Arm/Group | Placebo of Pradigastat (LCQ908) Regimen | 20 mg Pradigastat (LCQ908) Regimen | 40 mg Pradigastat (LCQ908) Regimen | Pradigastat (LCQ908) Regimen- From Study A2212
Started | 5 | 6 | 4 | 4
Completed | 0 | 0 | 0 | 0
Not Completed | 5 | 6 | 4 | 4
Not completed — Subject/guardian decision | 0 | 1 | 0 | 0
Not completed — Study terminated by sponsor | 5 | 5 | 4 | 3
Not completed — Physician Decision | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) - All subjects in the extension study who were in full analysis set in either study LCQ908A2212/NCT01146522 or LCQ908B2302/NCT01514461.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo of Pradigastat (LCQ908) Regimen | 20 mg Pradigastat (LCQ908) Regimen | 40 mg Pradigastat (LCQ908) Regimen | Pradigastat (LCQ908) Regimen- From Study A2212 | Total
Number analyzed (Participants) | 11 | 12 | 10 | 5 | 38
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.9 (10.22) | 44.1 (14.26) | 43.6 (84.53) | 52.2 (12.72) | 47.6 (11.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 2 | 3 | 16
  Male | 6 | 6 | 8 | 2 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Any Adverse Events, Serious Adverse Events and Death
Time Frame: 52 weeks
Population: Safety set (SAF) - All subjects who received at least one dose of study drug and had at least one post-baseline safety assessment in this extension study.
Measure: Number; unit: Participants
Groups:
- Placebo of Pradigastat (LCQ908) Regimen: Part A: Patients who were randomized to placebo in study CLCQ908B2302/NCT01514461. In current study, patients initiated at 10 mg/day. After at least 8 weeks of treatment with a dose, optional up-titration to the next possible dose was allowed. One down titration allowed from the highest dose attained.
- 20 mg Pradigastat (LCQ908) Regimen: Part A: Patients who were randomized to LCQ908 20 mg in study CLCQ908B2302/NCT01514461. In current study, patients initiated at LCQ908 10 mg/day. After at least 8 weeks of treatment with a dose, optional up-titration to the next possible dose was allowed. One down titration allowed from the highest dose attained.
- 40 mg Pradigastat (LCQ908) Regimen: Part A: Patients who were randomized to LCQ908 40 mg in study CLCQ908B2302/NCT01514461. In current study, patients initiated at LCQ908 10 mg/day. After at least 8 weeks of treatment with a dose, optional up-titration to the next possible dose was allowed. One down titration allowed from the highest dose attained.
- Pradigastat (LCQ908) Regimen- From Study A2212: Part A: Patients who were randomized to LCQ908 in study CLCQ908A2212/NCT01146522. In current study, patients initiated at LCQ908 10 mg/day. After at least 8 weeks of treatment with a dose, optional up-titration to the next possible dose was allowed. One down titration allowed from the highest dose attained.
Arm/Group | Placebo of Pradigastat (LCQ908) Regimen | 20 mg Pradigastat (LCQ908) Regimen | 40 mg Pradigastat (LCQ908) Regimen | Pradigastat (LCQ908) Regimen- From Study A2212
Number analyzed (Participants) | 11 | 12 | 10 | 5
Participants
  At least one Adverse Event (any) | 11 | 12 | 10 | 5
  At least one serious AE | 1 | 6 | 2 | 2
  Death | 0 | 0 | 0 | 0

2. Secondary Outcome: Changes From Baseline in Triglyceride Levels up to 52 Weeks
Description: Blood samples were collected for a fasting lipid panel, including total triglycerides. Lipid measurements were collected after a 12 hour (overnight) fast. The maintenance of effect was assessed on triglyceride levels during continued therapy with LCQ908 for up to 52 weeks. For patients from LCQ908 arm of study CLCQ908A2212, baseline was the assessment obtained at Week 0 of current study. For patients from study CLCQ908B2302, baseline is defined as the average of values taken Day -3 and Week 0 (randomization) in study CLCQ908B2302. The geometric mean for the percentage (%) change is calculated from back-transforming the mean of the log transformed ratio to baseline values: (exp(mean of the log-transformed ratio to baseline values) -1)*100.
Time Frame: Baseline, Week 12, 24 and 52
Population: Full analysis set (FAS) - All subjects in the extension study who were in FAS in either study LCQ908A2212 or LCQ908B2302. At each time point post-baseline, only patients with a value at both baseline and the post-dose time point are included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage change
Arm/Group | Placebo of Pradigastat (LCQ908) Regimen | 20 mg Pradigastat (LCQ908) Regimen | 40 mg Pradigastat (LCQ908) Regimen | Pradigastat (LCQ908) Regimen- From Study A2212
Number analyzed (Participants) | 11 | 12 | 10 | 5
percentage change
  Change in week 12 (n=10,11,10,5) | 1.63 (45.19) | -5.80 (66.10) | 43.94 (52.66) | -19.36 (42.82)
  change in week 24 (n=10,10,9,5) | -14.59 (52.33) | -36.19 (64.80) | 32.54 (87.83) | -26.05 (31.50)
  change in week 52 (n=9,8,9,5) | 16.46 (29.27) | -30.03 (78.52) | 92.15 (60.21) | -9.20 (43.34)

3. Secondary Outcome: Changes From Baseline in Cholesterol Levels up to 52 Weeks
Description: Blood samples were collected for a fasting lipid panel, including cholesterol level. Lipid measurements were collected after a 12 hour (overnight) fast. For patients from LCQ908 arm of study CLCQ908A2212, baseline was the assessment obtained at Week 0 of current study. For patients from study CLCQ908B2302, baseline is defined as the average of values taken Day -3 and Week 0 (randomization) in study CLCQ908B2302. The geometric mean for the percentage (%) change is calculated from back-transforming the mean of the log transformed ratio to baseline values: (exp(mean of the log-transformed ratio to baseline values) -1)*100.
Time Frame: Baseline, Week 12, 24 and 52
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage change
Arm/Group | Placebo of Pradigastat (LCQ908) Regimen | 20 mg Pradigastat (LCQ908) Regimen | 40 mg Pradigastat (LCQ908) Regimen | Pradigastat (LCQ908) Regimen- From Study A2212
Number analyzed (Participants) | 11 | 12 | 10 | 5
percentage change
  Change in week 12 (n=10,11,10,5) | -5.58 (36.38) | -4.76 (36.26) | 18.76 (31.54) | -10.42 (24.68)
  change in week 24 (n=10,10,9,5) | -10.54 (27.87) | -21.54 (24.98) | 7.45 (37.28) | -13.87 (25.64)
  change in week 52 (n=9,8,9,5) | 5.75 (17.51) | -13.76 (36.10) | 40.95 (34.10) | -6.84 (22.55)

4. Secondary Outcome: Changes From Baseline in HDL and Non HDL Cholesterol Levels up to 52 Weeks
Description: Blood samples were collected for a fasting lipid panel, including HDL and non HDL cholesterol level. Lipid measurements were collected after a 12 hour (overnight) fast. For patients from LCQ908 arm of study CLCQ908A2212, baseline was the assessment obtained at Week 0 of current study. For patients from study CLCQ908B2302, baseline is defined as the average of values taken Day -3 and Week 0 (randomization) in study CLCQ908B2302. The geometric mean for the percentage (%) change is calculated from back-transforming the mean of the log transformed ratio to baseline values: (exp(mean of the log-transformed ratio to baseline values) -1)*100.
Time Frame: Baseline, Week 12, 24 and 52
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage change
Arm/Group | Placebo of Pradigastat (LCQ908) Regimen | 20 mg Pradigastat (LCQ908) Regimen | 40 mg Pradigastat (LCQ908) Regimen | Pradigastat (LCQ908) Regimen- From Study A2212
Number analyzed (Participants) | 11 | 12 | 10 | 5
percentage change
  HDL: Change in week 12 (n=10,11,10,5) | -14.13 (30.08) | 3.37 (24.75) | -5.99 (22.19) | -7.09 (27.11)
  Non HDL: change in week 12 (n=10,11,10,5) | -5.37 (39.61) | -7.72 (42.40) | 20.70 (34.18) | -10.57 (26.16)
  HDL: change in week 24 (n=10,10,9,5) | -7.11 (19.41) | -1.83 (31.36) | 6.67 (22.19) | -15.60 (37.69)
  Non HDL: change in week 24 (n=10,10,9,5) | -11.29 (29.53) | -25.22 (31.49) | 7.17 (40.50) | -14.01 (28.04)
  HDL: change in week 52 (n=9,8,9,5) | -10.85 (19.78) | 8.11 (29.35) | -7.33 (27.63) | -21.41 (22.91)
  Non HDL: change in week 52 (n=9,8,9,5) | 8.06 (21.42) | -17.68 (42.65) | 45.25 (37.45) | -6.09 (24.59)

5. Secondary Outcome: Changes From Baseline in Glycerol Levels up to 52 Weeks
Description: Blood samples were collected for a fasting lipid panel, including glycerol level. Lipid measurements were collected after a 12 hour (overnight) fast. For patients from LCQ908 arm of study CLCQ908A2212, baseline was the assessment obtained at Week 0 of current study. For patients from study CLCQ908B2302, baseline is defined as the average of values taken Day -3 and Week 0 (randomization) in study CLCQ908B2302. The geometric mean for the percentage (%) change is calculated from back-transforming the mean of the log transformed ratio to baseline values: (exp(mean of the log-transformed ratio to baseline values) -1)*100.
Time Frame: Baseline, Week 12, 24 and 52
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage change
Arm/Group | Placebo of Pradigastat (LCQ908) Regimen | 20 mg Pradigastat (LCQ908) Regimen | 40 mg Pradigastat (LCQ908) Regimen | Pradigastat (LCQ908) Regimen- From Study A2212
Number analyzed (Participants) | 11 | 12 | 10 | 5
percentage change
  Change in week 12 (n=10,11,10,5) | -26.56 (72.88) | -15.50 (73.33) | 0.68 (75.40) | -46.83 (105.58)
  change in week 24 (n=10,10,9,5) | -40.00 (67.28) | -46.97 (62.46) | -36.26 (133.58) | -56.99 (96.06)
  change in week 52 (n=9,8,9,5) | -38.15 (70.10) | -31.96 (64.76) | -28.52 (101.85) | -37.02 (81.67)

6. Secondary Outcome: Changes From Baseline in Free Fatty Acid Levels up to 52 Weeks
Description: Blood samples were collected for a fasting lipid panel, including free fatty acid level. Lipid measurements were collected after a 12 hour (overnight) fast. For patients from LCQ908 arm of study CLCQ908A2212, baseline was the assessment obtained at Week 0 of current study. For patients from study CLCQ908B2302, baseline is defined as the average of values taken Day -3 and Week 0 (randomization) in study CLCQ908B2302. The geometric mean for the percentage (%) change is calculated from back-transforming the mean of the log transformed ratio to baseline values: (exp(mean of the log-transformed ratio to baseline values) -1)*100.
Time Frame: Baseline, Week 12, 24 and 52
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage change
Arm/Group | Placebo of Pradigastat (LCQ908) Regimen | 20 mg Pradigastat (LCQ908) Regimen | 40 mg Pradigastat (LCQ908) Regimen | Pradigastat (LCQ908) Regimen- From Study A2212
Number analyzed (Participants) | 11 | 12 | 10 | 5
percentage change
  Change in week 12 (n=10,11,10,5) | -23.11 (53.05) | -17.85 (62.48) | 53.09 (44.83) | -46.58 (128.38)
  change in week 24 (n=10,10,9,5) | -20.35 (80.16) | -30.44 (62.01) | 36.18 (64.97) | -42.74 (108.73)
  change in week 52 (n=9,8,9,5) | -16.99 (43.34) | -7.69 (54.21) | 79.15 (49.37) | -18.29 (104.77)

7. Secondary Outcome: Changes From Baseline in Apolipoprotein A1 Levels up to 52 Weeks
Description: Fasting blood samples were collected by direct venipuncture or an indwelling cannula to evaluate the drug effect on lipoprotein biomarkers such as Apolipoprotein A1. For patients from LCQ908 arm of study CLCQ908A2212, baseline was the assessment obtained at Week 0 of current study. For patients from study CLCQ908B2302, baseline is defined as the average of values taken Day -3 and Week 0 (randomization) in study CLCQ908B2302. The geometric mean for the percentage (%) change is calculated from back-transforming the mean of the log transformed ratio to baseline values: (exp(mean of the log-transformed ratio to baseline values) -1)*100.
Time Frame: Baseline, Week 12, 24 and 52
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage change
Arm/Group | Placebo of Pradigastat (LCQ908) Regimen | 20 mg Pradigastat (LCQ908) Regimen | 40 mg Pradigastat (LCQ908) Regimen | Pradigastat (LCQ908) Regimen- From Study A2212
Number analyzed (Participants) | 11 | 12 | 10 | 5
percentage change
  Change in week 12 (n=11,11,10,5) | -3.24 (23.82) | 2.55 (15.09) | 6.58 (17.04) | 2.95 (33.54)
  change in week 24 (n=10,10,10,5) | 4.80 (14.16) | 1.41 (17.45) | 5.57 (25.69) | 5.11 (28.49)
  change in week 52 (n=10,8,9,5) | 4.51 (19.21) | 10.01 (16.28) | 4.43 (19.34) | -0.82 (16.79)

8. Secondary Outcome: Changes From Baseline in Apolipoprotein B-48 Levels up to 52 Weeks
Description: Fasting blood samples were collected by direct venipuncture or an indwelling cannula to evaluate the drug effect on lipoprotein biomarkers such as Apolipoprotein B-48. For patients from LCQ908 arm of study CLCQ908A2212, baseline was the assessment obtained at Week 0 of current study. For patients from study CLCQ908B2302, baseline is defined as the average of values taken Day -3 and Week 0 (randomization) in study CLCQ908B2302. The geometric mean for the percentage (%) change is calculated from back-transforming the mean of the log transformed ratio to baseline values: (exp(mean of the log-transformed ratio to baseline values) -1)*100.
Time Frame: Baseline, Week 12, 24 and 52
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage change
Arm/Group | Placebo of Pradigastat (LCQ908) Regimen | 20 mg Pradigastat (LCQ908) Regimen | 40 mg Pradigastat (LCQ908) Regimen | Pradigastat (LCQ908) Regimen- From Study A2212
Number analyzed (Participants) | 11 | 12 | 10 | 5
percentage change
  Change in week 12 (n=11,11,10,5) | -4.03 (79.87) | 33.24 (79.20) | 109.67 (52.50) | -30.03 (61.78)
  change in week 24 (n=10,10,10,5) | 9.13 (30.79) | -10.23 (58.91) | 105.52 (71.45) | -35.04 (31.11)
  change in week 52 (n=10,8,9,5) | 56.25 (57.65) | -22.63 (107.21) | 135.33 (71.11) | 27.75 (57.77)

9. Secondary Outcome: Changes From Baseline in Apolipoprotein B-100 Levels up to 52 Weeks
Description: Fasting blood samples were collected by direct venipuncture or an indwelling cannula to evaluate the drug effect on lipoprotein biomarkers such as Apolipoprotein B-100. For patients from LCQ908 arm of study CLCQ908A2212, baseline was the assessment obtained at Week 0 of current study. For patients from study CLCQ908B2302, baseline is defined as the average of values taken Day -3 and Week 0 (randomization) in study CLCQ908B2302. The geometric mean for the percentage (%) change is calculated from back-transforming the mean of the log transformed ratio to baseline values: (exp(mean of the log-transformed ratio to baseline values) -1)*100.
Time Frame: Baseline, Week 12, 24 and 52
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage change
Arm/Group | Placebo of Pradigastat (LCQ908) Regimen | 20 mg Pradigastat (LCQ908) Regimen | 40 mg Pradigastat (LCQ908) Regimen | Pradigastat (LCQ908) Regimen- From Study A2212
Number analyzed (Participants) | 11 | 12 | 10 | 5
percentage change
  Change in week 12 (n=9,11,9,5) | -15.75 (41.50) | 15.10 (58.53) | -8.34 (32.73) | 3.33 (32.46)
  change in week 24 (n=10,9,10,5) | -2.75 (63.10) | 21.33 (38.76) | -18.28 (52.94) | 11.68 (43.73)
  change in week 52 (n=10,7,9,5) | -12.52 (44.16) | 25.39 (36.77) | -10.73 (37.20) | 10.02 (39.08)

ADVERSE EVENTS:
Groups:
- Part A-placebo of Pradigastat (LCQ908) Regimen: Part A: Patients who were randomized to placebo in study CLCQ908B2302/NCT01514461. In current study, patients initiated at 10 mg/day. After at least 8 weeks of treatment with a dose, optional up-titration to the next possible dose was allowed. One down titration allowed from the highest dose attained.
- Part A-20mg Pradigastat (LCQ908) Regimen: Part A: Patients who were randomized to LCQ908 20 mg in study CLCQ908B2302/NCT01514461. In current study, patients initiated at LCQ908 10 mg/day. After at least 8 weeks of treatment with a dose, optional up-titration to the next possible dose was allowed. One down titration allowed from the highest dose attained.
- Part A-40mg Pradigastat (LCQ908) Regimen: Part A: Patients who were randomized to LCQ908 40 mg in study CLCQ908B2302/NCT01514461. In current study, patients initiated at LCQ908 10 mg/day. After at least 8 weeks of treatment with a dose, optional up-titration to the next possible dose was allowed. One down titration allowed from the highest dose attained.
- Part A: Pradigastat (LCQ908) Regimen- From Study A2212: Part A: Patients who were randomized to LCQ908 in study CLCQ908A2212/NCT01146522. In current study, patients initiated at LCQ908 10 mg/day. After at least 8 weeks of treatment with a dose, optional up-titration to the next possible dose was allowed. One down titration allowed from the highest dose attained.
- Part B-placebo of Pradigastat (LCQ908) Regimen; Part B-20mg Pradigastat (LCQ908) Regimen; Part B- Pradigastat (LCQ908) Regimen- From Study A2212; Part B-40 mg Pradigastat (LCQ908): Part B: Patients who consented to take part in the Part B continued their treatment at the same dose as they took when they completed Part A. LCQ908 treatment could be titrated (within the dose range 10 mg to 40 mg) at the investigators discretion and based on individual patients' tolerance and safety profile.
Arm/Group | Part A-placebo of Pradigastat (LCQ908) Regimen | Part A-20mg Pradigastat (LCQ908) Regimen | Part A-40mg Pradigastat (LCQ908) Regimen | Part A: Pradigastat (LCQ908) Regimen- From Study A2212 | Part B-placebo of Pradigastat (LCQ908) Regimen | Part B-20mg Pradigastat (LCQ908) Regimen | Part B- Pradigastat (LCQ908) Regimen- From Study A2212 | Part B-40 mg Pradigastat (LCQ908)
Serious Adverse Events (participants affected / at risk) | 1/11 | 6/12 | 2/10 | 2/5 | 0/5 | 0/6 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 11/11 | 12/12 | 10/10 | 5/5 | 4/5 | 3/6 | 3/4 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A-placebo of Pradigastat (LCQ908) Regimen (N=11) | Part A-20mg Pradigastat (LCQ908) Regimen (N=12) | Part A-40mg Pradigastat (LCQ908) Regimen (N=10) | Part A: Pradigastat (LCQ908) Regimen- From Study A2212 (N=5) | Part B-placebo of Pradigastat (LCQ908) Regimen (N=5) | Part B-20mg Pradigastat (LCQ908) Regimen (N=6) | Part B- Pradigastat (LCQ908) Regimen- From Study A2212 (N=4) | Part B-40 mg Pradigastat (LCQ908) (N=4)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
CORONARY ARTERY STENOSIS (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
PANCREATITIS (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
GASTROENTERITIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
MALNUTRITION (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A-placebo of Pradigastat (LCQ908) Regimen (N=11) | Part A-20mg Pradigastat (LCQ908) Regimen (N=12) | Part A-40mg Pradigastat (LCQ908) Regimen (N=10) | Part A: Pradigastat (LCQ908) Regimen- From Study A2212 (N=5) | Part B-placebo of Pradigastat (LCQ908) Regimen (N=5) | Part B-20mg Pradigastat (LCQ908) Regimen (N=6) | Part B- Pradigastat (LCQ908) Regimen- From Study A2212 (N=4) | Part B-40 mg Pradigastat (LCQ908) (N=4)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
CARDIAC FAILURE (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
ABNORMAL PALMAR/PLANTAR CREASES (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
EAR PAIN (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
VERTIGO POSITIONAL (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 0 | 1 | 1 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 8 | 11 | 5 | 4 | 2 | 1 | 3 | 0
DYSPEPSIA (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
FAECAL INCONTINENCE (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
FOOD POISONING (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
GASTRITIS (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 2 | 4 | 3 | 2 | 2 | 2 | 0 | 0
PANCREATITIS (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
STEATORRHOEA (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
TONGUE CYST (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
VOMITING (Gastrointestinal disorders) | 1 | 2 | 1 | 1 | 1 | 0 | 0 | 0
FATIGUE (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
THIRST (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
VESSEL PUNCTURE SITE INDURATION (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
BRONCHITIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
CYSTITIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
GASTROENTERITIS (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
INFLUENZA (Infections and infestations) | 6 | 2 | 2 | 0 | 0 | 0 | 0 | 0
LUNG INFECTION (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
NASOPHARYNGITIS (Infections and infestations) | 4 | 4 | 0 | 1 | 2 | 1 | 0 | 0
PNEUMONIA (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
POST PROCEDURAL INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
SINUSITIS (Infections and infestations) | 1 | 2 | 1 | 1 | 1 | 0 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
VAGINAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
CONTUSION (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
FALL (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
LIGAMENT RUPTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
POST PROCEDURAL INFLAMMATION (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
WOUND (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
CARDIAC MURMUR (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
CAROTID BRUIT (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
WEIGHT DECREASED (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
GOUT (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
VITAMIN B COMPLEX DEFICIENCY (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
TENDONITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
APHONIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
DIZZINESS (Nervous system disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0
HEADACHE (Nervous system disorders) | 1 | 2 | 2 | 1 | 0 | 0 | 0 | 0
MIGRAINE (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
PARAESTHESIA (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
RESTLESS LEGS SYNDROME (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
SCIATICA (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
SYNCOPE (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
AGITATION (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
DEPRESSED MOOD (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
INSOMNIA (Psychiatric disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
STRESS (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
DYSMENORRHOEA (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
PREMATURE MENOPAUSE (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
PHARYNGEAL INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
PSORIASIS (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
XANTHOMA (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
AORTIC ANEURYSM (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
HOT FLUSH (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
HYPERTENSION (Vascular disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
As the anticipated benefit from the continued participation of patients in 18 month extension (Part B) was not supported by results of the December 2014 interim analysis, Novartis decided to terminate the Part B to be effective as of May 31, 2015.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.